CLINICAL TRIAL: NCT01707277
Title: The Effects of Inspiratory Muscle Training in Patients With Heart Failure With Preserved Ejection Fraction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación para la Investigación del Hospital Clínico de Valencia (Other)
Collaborators: University of Valencia (Other)
Responsible Party: Principal Investigator, Julio Nuñez, MD, PhD, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EMI
Record Dates: First submitted 2012-10-09; First posted 2012-10-16 (Estimated); Last update posted 2016-02-04 (Estimated); Status verified 2016-02

CONDITIONS: Heart Failure
Keywords: Heart failure with preserved ejection fraction; Inspiratory muscle training; Exercise capacity
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Inspiratory muscle training (Experimental): Inspiratory muscle training for improving maximum inspiratory pressure plus phrmacological treatment Pharmacological treatment (usual care)
  Interventions: Other: Inspiratory muscle training; Other: Usual care
- Usual care (Active Comparator): Pharmacological treatment
  Interventions: Other: Usual care

INTERVENTIONS:
Other: Inspiratory muscle training — Patients were instructed to train at home twice daily for 20 minutes each session during 12 weeks with a threshold inspiratory muscle trainer (Threshold IMT®, Respironics Inc.). All of them were trained under the supervision of a physiotherapist and educated to maintain diaphragmatic breathing during training. The subjects started breathing at a resistance equal to 25-30% of their maximum inspiratory pressure for 1 week.
  Arms: Inspiratory muscle training
Other: Usual care — Usual pahramacological treatment

SUMMARY:
Previous studies have evaluated the effects of inspiratory muscle training in patiens with heart failure and reduced ejection fraction; nevertheless,no evidence endorse the therapeutic role of inspiratory muscle training in patients with heart failure and preserved ejection fraction. The investigators sought to evaluate whether 12-week inspiratory muscle training improves exercise capacity (peak exercise oxygen uptake and 6-minutes walk test), as well as left ventricular diastolic function, serum biomarkers and quality of life (Minnesota Living With Heart Failure Questionnaire) in patients with heart failure with preserved ejection fraction and non-reduced inspiratory muscle strength.

ELIGIBILITY:
Inclusion Criteria:

* a) previous history of symptomatic heart failure (New York Heart Association [NYHA] functional class ≥II)
* b) evidence of normal left ventricular ejection fraction, defined by an ejection fraction >0.50 and an end-diastolic diameter <60 mm by 2D echocardiography
* c) relevant structural heart disease (left ventricle hypertrophy/left atrial enlargement) and/or diastolic dysfunction estimated by 2D echocardiography
* d) clinical stability, including no admissions in the past 30 days

Exclusion Criteria:

* a) Patients unable to perform a valid baseline exercise test.
* b) Unstable angina, myocardial infarction or cardiac surgery within the previous three months.
* c)Known chronic metabolic, orthopedic, infectious disease or previous pulmonary disease;
* d)Treatment with steroids, hormones, or cancer chemotherapy;
* e)Reduced maximal inspiratory pressure according to age and sex;
* f)Active smokers
* g)Acute decompensation;
* h)Other comorbidity with an expectancy of life less than one year

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2011-03; Primary Completion 2012-01 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Changes in exercise capacity parameters at 12-weeks. | 12 weeks
  Exercise parameters: peak exercise oxygen uptake (peak VO2), 6-minutes walk test

SECONDARY OUTCOMES:
Changes in 12-week quality of life, biomarkers related to the severity and parameters of left ventricular diastolic function. | 12 weeks
  Quality of life: Minnesota Living With Heart Failure Questionnaire. Biomarkers: plasma natriuretic peptides, estimaated glomerular filtration rate, antigen carbohydrate 125.
  Diastolic function: E/e´.

CONTACTS AND LOCATIONS:
Overall Officials: Julio Núñez, MD, Principal Investigator — Hospital Clínico Universitario de Valencia
Locations (1):
- Hospital Clínico Universitario, Valencia, Valencia, Spain

REFERENCES:
- [Background] Lin SJ, McElfresh J, Hall B, Bloom R, Farrell K. Inspiratory muscle training in patients with heart failure: a systematic review. Cardiopulm Phys Ther J. 2012 Sep;23(3):29-36. PMID 22993500
- [Derived] Diaz-Buschmann I, Jaureguizar KV, Calero MJ, Aquino RS. Programming exercise intensity in patients on beta-blocker treatment: the importance of choosing an appropriate method. Eur J Prev Cardiol. 2014 Dec;21(12):1474-80. doi: 10.1177/2047487313500214. Epub 2013 Aug 5. PMID 23918838
- [Derived] Palau P, Dominguez E, Nunez E, Schmid JP, Vergara P, Ramon JM, Mascarell B, Sanchis J, Chorro FJ, Nunez J. Effects of inspiratory muscle training in patients with heart failure with preserved ejection fraction. Eur J Prev Cardiol. 2014 Dec;21(12):1465-73. doi: 10.1177/2047487313498832. Epub 2013 Jul 17. PMID 23864363